CLINICAL TRIAL: NCT01267526
Title: "Easypod™ Connect Registry": A Canadian, Multi-centre, Observational Registry to Study Adherence and Long Term Outcomes of SAIZEN® in Pediatric Subjects Using Easypod™ Auto-injector
Brief Title: A Canadian, Multi-centre, Observational Registry to Study Adherence and Long Term Outcomes of Therapy in Pediatric Subjects Using SAIZEN® Via Easypod™ Auto-injector for Growth Hormone Treatment
Acronym: ECOS CAN
Status: Completed | Type: Observational
Sponsor: Merck KGaA, Darmstadt, Germany (Industry)
Collaborators: EMD Serono, a division of EMD Inc., Canada (Industry)
Responsible Party: Sponsor
Other Study IDs: EMR200104-517
Record Dates: First submitted 2010-12-27; First posted 2010-12-28 (Estimated); Last update posted 2017-12-26 (Actual); Status verified 2017-12

CONDITIONS: Growth Disorders
Keywords: Growth disorders; Saizen; Easypod; Growth hormone; Pediatric subject
MeSH Terms: conditions — Growth Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: Easypod™ — Saizen (Somatotropin) administered by easypod™ as defined in SAIZEN® Canadian Product Monograph
  Other Names: Saizen; Somatropin

SUMMARY:
This is a Canadian, Multicentre, Observational Registry to study Adherence and Long Term Outcomes of Therapy in paediatric subjects using Easypod™ electromechanical device for growth hormone treatment from hospital and to assess the level of adherence of subject receiving SAIZEN® via Easypod™ .

DETAILED DESCRIPTION:
Subjects will be enrolled in a multicenter, longitudinal observational registry. Parents/subjects will provide their Informed Consent/assent to upload their data for populationbased analyses and optionally to adhere to a patient adherence support program designed to improve their adherence and, ultimately, clinical outcomes. Adherence data will be primarily derived from the Easypod™ device combined with physician data entry of outcome measures. Data will be collected retrospectively and prospectively. This will allow the establishment of adherence profiles and explore the hypothesis that patient adherence support programs improve adherence and subsequent clinical outcomes. Collected data will be also analyzed in a multinational pooled analysis of comparable national studies.

Primary Objective:

- To assess the level of adherence of subjects prescribed SAIZEN® via easypod™

Secondary Objectives:

* To describe the impact of adherence on clinical outcomes for subject prescribed SAIZEN via easypod™
* To identify adherence subject profiling

ELIGIBILITY:
Inclusion Criteria:

* Prescribed SAIZEN® via the easypod™ auto-injector (SAIZEN® Health Canadian approved indications: Growth Hormone Insufficiency or Deficiency, Turner's Syndrome, Chronic Renal Failure, Small for Gestational Age
* Under 18 years of age, or over 18 without fusion of growth plates
* Parent's or legal guardian's written informed consent, given before entering data into the registry, with the understanding that the subject or parent/legal guardian may withdraw consent at any time without prejudice to future medical care. If the child is old enough to read and write, a separate assent form will be given as defined by Health Canada regulations. Adult consent is defined at 18+ in the province of Quebec, 16+ in the remainder of Canada.

Exclusion Criteria:

* Subjects taking growth hormone in whom growth plates have fused (i.e. for taking growth hormone for its metabolic effects)
* Contra-indications to SAIZEN® as defined in SAIZEN® Canadian Product Monograph.
* Use of an investigational drug or participation in another interventional clinical study

Ages: 2 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Pediatric subjects 18 and under who are prescribed SAIZEN® (Health Canada approved indications) using the easypod™ auto-injector.
Sampling Method: Non-Probability Sample
Enrollment: 205 (Actual)
Dates: Start 2011-05-31 (Actual); Primary Completion 2015-12-31 (Actual); Study Completion 2015-12-31 (Actual)

PRIMARY OUTCOMES:
Mean percent of adherence by subject over a period of time | At least 6 months and up to 5 years
  Adherence will be defined as 86 percent adherent at one year based on prescribed therapy.

SECONDARY OUTCOMES:
Correlation of adherence and growth outcome after each year of SAIZEN® treatment with easypod™ | At least 6 months and up to 5 years
  Correlation of adherence and growth outcome (height velocity (HV), height velocity-standard deviation score (HV-SDS), height, change in height (height SDS) after each year of SAIZEN® treatment with easypod™
Subject adherence profile based on age, gender, indication, self-injection or not, time on treatment | At least 6 months and up to 5 years
Impact of patient adherence support programme on adherence and outcomes for subjects using easypod™ | At least 6 months and up to 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Medical Responsible, Study Director — EMD Serono, a division of EMD Inc., Canada
Locations (9):
- Canada (9):
  - Merck Serono Research Site, Calgary, Alberta
  - Merck Serono Research Site, Edmonton, Alberta
  - Merck Serono Research Site, North Vancouver, British Columbia
  - Merck Serono Research Site, Vancouver, British Columbia
  - Merck Serono Research Site, Hamilton, Ontario
  - Merck Serono Research Site, London, Ontario
  - Merck Serono Research Site, Toronto, Ontario
  - Merck Serono Research Site, Montreal, Quebec
  - Merck Serono Research Site, Sherbrooke, Quebec

REFERENCES:
- [Result] Koledova, E. et al. (2017) Analysis of results from the global, 5-year Easypod™ Connect Observational Study (ECOS) study in children with growth disorders. 10th International Meeting for Pediatric Endocrinology; 2017 Sep 14-17; Washington, DC.
- [Result] Wit, JM. et al. (2017) Effect of adherence on the 2-year growth response to growth hormone treatment in prepubertal children with idiopathic isolated growth hormone deficiency participating in the EasypodTM Connect Observational Study (ECOS). 10th International Meeting of Paediatric Endocrinology; 2017 Sep 14-17; Washington, DC.